CLINICAL TRIAL: NCT03583996
Title: The HepQuant SHUNT Liver Diagnostic Kit for Likelihood of Large Esophageal Varices: The SHUNT-V Study
Brief Title: The SHUNT-V Study for Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HepQuant, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HQ-US-SHUNT-1801
Record Dates: First submitted 2018-04-20; First posted 2018-07-12 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Intervention Model Description: All subjects receive HepQuant SHUNT test and DSI measurement prior to a standard of care (SOC) EGD, to be done within 42 days of the SHUNT test. HepQuant SHUNT is a combination product where 24-13C-cholic acid (13C cholate) 20mg is administered intravenously once for each test and 2,2,4,4-D4-cholic acid (d4 cholate) 40mg is administered once orally for each test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open Label (Experimental): All subjects receive HepQuant SHUNT Liver Diagnostic Test within 42 days of the scheduled EGD. Test includes 20mg of 13C Cholate mixed with Albumin via IV push, and 40mg of d4 Cholate mixed with juice orally, both doses given simultaneously one time.
  Interventions: Combination Product: HepQuant SHUNT Liver Diagnostic Test

INTERVENTIONS:
Combination Product: HepQuant SHUNT Liver Diagnostic Test — One time testing using the HepQuant SHUNT Liver Diagnostic Test kit (the combination product) in subjects with CLD and undergoing a standard of care EGD. The SHUNT test will be completed prior to the EGD. Each subject will receive an IV push dose of 13C Cholate mixed with Albumin simultaneously with an oral dose of d4 Cholate

SUMMARY:
The purpose of this study is to validate the Disease Severity Index (DSI) from the HepQuant SHUNT Liver Diagnostic Kit (Test) for likelihood of large esophageal varices.

DETAILED DESCRIPTION:
The purpose of this study is to validate the Disease Severity Index (DSI) from the HepQuant SHUNT Liver Diagnostic Kit (Test) for likelihood of large esophageal varices. The Hepatitis C Antiviral Long-term Treatment against Cirrhosis (HALT-C) Trial training dataset demonstrated that the DSI 18.3 had sensitivity 95%, specificity 54%, positive predictive value (PPV) 19%, negative predictive value (NPV) >99%, negative likelihood ratio (NLR) 0.09, and positive likelihood ratio (PLR) 2.09 for large varices. To validate DSI 18.3 as a cutoff for large varices, we will enroll 420 subjects with chronic liver disease (CLD) of mixed etiologies from 15 to 25 US clinical centers (CLD Validation dataset). The target prevalence of large varices is ≥20%. Each subject will have been scheduled for an esophago-gastro-duodenoscopy (EGD) as part of their standard of care for either variceal or non-variceal indications. Enrolled subjects will undergo standard clinical assessment, laboratory tests, and the HepQuant SHUNT Test. The EGD will be performed within 6 weeks following the HepQuant SHUNT Test. The relationship of DSI to large varices will be analyzed by univariate and multivariate logistic regression analyses, area under the receiver operating characteristic curve (AUROC), and linear and nonlinear regression and correlation coefficients. Diagnostic performance of the DSI cutoff will be defined in the CLD Validation dataset and validated for likelihood of large esophageal varices. The validated DSI cutoff will identify subjects who are either unlikely or likely to have large esophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* Ability to have a peripheral venous catheter for administration of the 13C cholate
* Ability to take the oral dose of d4-cholate
* Ability to hold morning doses of medications for the 90-minute duration of the HepQuant SHUNT Test
* Meets the protocol defined criteria for CLD in addition to having the diagnoses of CLD for >6 months
* Is scheduled, or in the process of being scheduled, for a standard of care EGD

Exclusion Criteria:

* Unable to give informed consent
* Unable to obtain venous access for administration of intravenous cholate
* Unable to absorb orally-administered cholate
* Known hypersensitivity to human serum albumin
* Known hypersensitivity to any of the components of the HepQuant SHUNT Liver Diagnostic Kit
* Acute hepatitis or Acute Liver Failure
* Acute drug-induced liver disease (DILI)
* Noncirrhotic causes for portal hypertension and varices
* Ongoing active alcoholic hepatitis
* Child-Pugh class C defined by Child-Pugh score 10 or higher
* Dialysis
* Active infection or febrile illness within the last month
* Documented history of esophageal or gastric variceal hemorrhage
* Documented history of treatment of esophageal varices
* Documented history of endoscopic findings of large esophageal varices
* Hepatocellular carcinoma beyond Milan or University of California, San Francisco (UCSF) criteria
* Thrombosis of main portal vein
* Liver transplant recipient
* Pregnancy
* Women who are breast-feeding
* Serious intercurrent medical or surgical illness, such as acute myocardial infarction, acute cerebral hemorrhage, sepsis, or other immediate life-threatening illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2022-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Everson, MD, Study Director — HepQuant, LLC
Locations (26):
- United States (26):
  - Arizona Liver Health, Chandler, Arizona
  - Southern CA Research Center, Coronado, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - Peak Gastroenterlogy Associates, Colorado Springs, Colorado
  - Nature Coast Clinical Research, Inverness, Florida
  - Mayo Clinic, Jacksonville, Jacksonville, Florida
  - Accel Research Sites, Orange City, Florida
  - Gastroenterology Associates of Pensacola, Pensacola, Florida
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Digestive Disease Associates, Catonsville, Maryland
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - St Louis University, St Louis, Missouri
  - Lucas Research (Diabetes & Endocrinology Consultants, PC), Morehead City, North Carolina
  - PMG Research, Winston-Salem, North Carolina
  - Univ of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Ralph H Johnson Veterans Affairs Medical Center, Charleston, South Carolina
  - Methodist Dallas Liver Center, Dallas, Texas
  - Baylor, Scott & White, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Intermountain Healthcare, Murray, Utah
  - Bon Secours, Newport News, Newport News, Virginia
  - Bon Secours, Richmond, Richmond, Virginia
  - Gastroenterology Consultants of SW VA, Roanoke, Virginia
  - University of WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiffman M, Reddy KR, Leise MD, Qureshi K, Smith AD, Helmke S, Kittelson J, McRae MP, Imperial JC, Everson GT; SHUNT-V Investigators. Cholate Shunt, Oral Cholate Challenge and Endoscopic Lesions of Portal Hypertension: The SHUNT-V Study. Aliment Pharmacol Ther. 2025 Jan;61(1):75-87. doi: 10.1111/apt.18386. Epub 2024 Nov 10. PMID 39523681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 367 subjects were screened for the study.
Pre-assignment Details: A total of 306 subjects were enrolled in the study. For the analyses of all primary, secondary, and exploratory endpoints, only subjects who completed the HepQuant SHUNT Test and esophagogastroduodenoscopy (EGD) examination (N=280) were considered.
Groups:
- Open Label: All subjects receive HepQuant SHUNT Liver Diagnostic Test within 42 days of the scheduled EGD. Test includes 20mg of 24-13C-cholic acid (13C cholate) mixed with Albumin via IV push, and 40mg of 2,2,4,4-D4-cholic acid (d4 cholate) mixed with juice orally, both doses given simultaneously one time.
  HepQuant SHUNT Liver Diagnostic Test: One time testing using the HepQuant SHUNT Liver Diagnostic Test kit (the combination product) in subjects with chronic liver disease (CLD) and undergoing a standard of care EGD. The SHUNT test was completed prior to the EGD. Each subject received an IV push dose of 13C Cholate mixed with Albumin simultaneously with an oral dose of d4 Cholate.
Period: Overall Study
Arm/Group | Open Label
Started | 280
Completed | 280
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Label: All subjects receive HepQuant SHUNT Liver Diagnostic Test within 42 days of the scheduled EGD. Test includes 20mg of 13C Cholate mixed with Albumin via IV push, and 40mg of d4 Cholate mixed with juice orally, both doses given simultaneously one time.
  HepQuant SHUNT Liver Diagnostic Test: One time testing using the HepQuant SHUNT Liver Diagnostic Test kit (the combination product) in subjects with CLD and undergoing a standard of care EGD. The SHUNT test was completed prior to the EGD. Each subject received an IV push dose of 13C Cholate mixed with Albumin simultaneously with an oral dose of d4 Cholate.
Arm/Group | Open Label
Number analyzed (Participants) | 280
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at informed consent
  years | 60.8 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140
  Male | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 1
  Race: Black or African American | 14
  Race: Native Hawaiian or other Pacific Islander | 0
  Race: White | 257
  Race: Other | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 44
  Ethnicity: Not Hispanic or Latino | 236
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Incomplete data entry
  kg/m^2
    number analyzed (Participants) | 278
    (all) | 33.48 (7.865)
Child-Pugh Score [Mean (Standard Deviation); unit: units on a scale] — The Child-Pugh score predicts mortality in patients with cirrhosis. The scale represents the severity of cirrhosis in three classes: Child-Pugh A, 5 to 6 points (well-compensated disease); Child-Pugh B, 7 to 9 points (significant functional impairment); Child-Pugh C, 10 to 15 points (decompensated disease). Population: Incomplete data entry
  units on a scale
    number analyzed (Participants) | 277
    (all) | 5.4 (0.84)
MELD Score [Mean (Standard Deviation); unit: units on a scale] — The Model for End-Stage Liver Disease (MELD) score is a numerical scale that estimates the survival probability during the next three months in patients with end-stage liver disease based on international normalized ratio (INR), serum total bilirubin, and serum creatinine. The MELD score ranges from 6 to 40. Higher values correspond to higher mortality risk. Population: Incomplete data entry
  units on a scale
    number analyzed (Participants) | 264
    (all) | 8.2 (2.66)

OUTCOME MEASURES:

1. Primary Outcome: Disease Severity Index (DSI) Less Than/Equal to 18.3 to Rule Out Large Varices
Description: The primary objective of this study is to measure the subjects' liver function using DSI ≤18.3 for those that are not likely to have large esophageal varices.
Time Frame: 1 day
Population: Of the 280 subjects who completed the HepQuant SHUNT Test and EGD examination, 275 had both HepQuant SHUNT Test and EGD results.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 275
Participants
  Large varices and DSI > 18.3 | 33
  Large varices and DSI <= 18.3 | 3
  No large varices and DSI > 18.3 | 171
  No large varices and DSI <= 18.3 | 68
Statistical Analysis 1: Comparison: Open Label; The performance goal for validation of DSI ≤18.3 was the upper limit of the confidence interval (CI) for negative likelihood ratio (NLR) to rule out an NLR of >0.52. For the null and alternate hypotheses, the upper limit of the 95% CI was NLR >0.52 and the upper limit of the 95% CI was NLR <=0.52, respectively. The confidence level for the CI was adjusted to maintain a 1-sided type I error rate of 0.025; Test type: Other; Negative Likelihood Ratio (NLR) = 0.293, 95% CI 2-sided [0.097 to 0.882]
Statistical Analysis 2: Comparison: Open Label; The performance goal for validation of DSI <= 18.3 was the observed sensitivity must have been >0.85. The confidence level for the confidence interval (CI) was adjusted to maintain a 1-sided type I error rate of 0.025; Test type: Other; Sensitivity = 0.917, 95% CI 2-sided [0.775 to 0.982]

2. Secondary Outcome: DSI and Probability of Large Esophageal Varices
Description: Logistic regression analysis of DSI as predictor of large varices
Time Frame: 1 day
Population: Of the 280 subjects who had the HepQuant SHUNT Test and EGD examination, 275 subjects had both HepQuant SHUNT Test and EGD.
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label
Number analyzed (Participants) | 275
Participants
  Large varices and DSI > 18.3 | 33
  Large varices and DSI <= 18.3 | 3
  No large varices and DSI > 18.3 | 171
  No large varices and DSI <= 18.3 | 68
Statistical Analysis 1: Comparison: Open Label; Test type: Other; p < 0.0001, Regression, Logistic — The odds ratio was for a 1-unit increase in DSI based on continuous DSI; Unadjusted (no covariates); Odds Ratio (OR) = 1.094, 95% CI 2-sided [1.047 to 1.143]
Statistical Analysis 2: Comparison: Open Label; Test type: Other; p < 0.0001, Regression, Logistic; Adjusted for demographic covariates, including age, race, sex, BMI, and ethnicity; Odds Ratio (OR) = 1.109, 95% CI 2-sided [1.058 to 1.163]
Statistical Analysis 3: Comparison: Open Label; Test type: Other; p < 0.001, Regression, Logistic; Adjusted for severity of liver disease covariates, compensated cirrhosis (CP class A); Odds Ratio (OR) = 1.092, 95% CI 2-sided [1.041 to 1.145]
Statistical Analysis 4: Comparison: Open Label; Test type: Other; p < 0.001, Regression, Logistic; Adjusted for severity of liver disease covariates, decompensated cirrhosis (CP class B); Odds Ratio (OR) = 1.089, 95% CI 2-sided [1.038 to 1.142]

ADVERSE EVENTS:
Time Frame: Information regarding adverse events (AE) and/or serious adverse events (SAE) were recorded during Visit 2 (HepQuant SHUNT Test Administration, <=28 days after enrollment) and Visit 3 (Post-Test Follow-up, 2 to 30 days after Visit 2). AEs and SAEs related to the performance of the EGD were recorded (note: findings of the EGD were NOT recorded as AEs).
Description: AEs/SAEs had their relationship to HepQuant SHUNT Liver Diagnostic Kit assessed by the clinician who examines and evaluates the participant based on temporal relationship and clinical judgment. Only 11 of the AEs below were related to HepQuant SHUNT test, and none of the intervention-related AEs were serious. Note: there were 297 subjects in the Safety Set which is different from the number of subjects that completed the study. All subjects in the Safety Set underwent the HepQuant SHUNT test.
Arm/Group | Open Label
All-Cause Mortality (participants affected / at risk) | 1/297
Serious Adverse Events (participants affected / at risk) | 5/297
Other Adverse Events (participants affected / at risk) | 40/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=297)
Coronary Artery Disease (Cardiac disorders) | 1 (1) — Moderate AE of coronary artery disease. The AE was an SAE and was considered unexpected and not related to the HepQuant SHUNT Liver Diagnostic Kit. The subject recovered from the AE but discontinued from the study because of the AE.
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Severe AE of pleural effusion. The AE was an SAE and was considered expected and not related to the HepQuant SHUNT Liver Diagnostic Kit. The subject recovered from the AE but discontinued from the study because of the AE.
Peritonitis Bacterial (Infections and infestations) | 1 (1) — Severe AEs of peritonitis bacterial and septic shock. The AEs were considered SAEs and were considered expected and not related to the HepQuant SHUNT Liver Diagnostic Kit. The subject died and was discontinued from the study because of the AEs.
Septic Shock (Infections and infestations) | 1 (1) — Severe AEs of peritonitis bacterial and septic shock. The AEs were considered SAEs and were considered expected and not related to the HepQuant SHUNT Liver Diagnostic Kit. The subject died and was discontinued from the study because of the AEs.
Hyperosmolar State (Metabolism and nutrition disorders) | 1 (1) — Moderate AE of hyperosmolar state. The AE of hyperosmolar state was an SAE and was considered unexpected and not related to the HepQuant SHUNT liver Diagnostic Kit. The subject recovered from the AE.
Metabolic Encephalopathy (Nervous system disorders) | 1 (1) — Moderate AE of metabolic encephalopathy. The AE of metabolic encephalopathy was an SAE and considered unexpected and not related to the HepQuant SHUNT Liver Diagnostic Kit. The subject recovered from the AE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label (N=297)
Infusion site bruising (General disorders) | 5 (8) — Related to HepQuant SHUNT Liver Diagnostic Kit
Catheter site bruise (General disorders) | 3 (3) — Related to HepQuant SHUNT Liver Diagnostic Kit
Infusion site pain (General disorders) | 1 (1) — Related to HepQuant SHUNT Liver Diagnostic Kit
Contusion (Injury, poisoning and procedural complications) | 2 (2) — One event in one affected subject was determined to be related to HepQuant SHUNT Liver Diagnostic Kit
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) — One event in one affected subject was determined to be related to HepQuant SHUNT Liver Diagnostic Kit
Diarrhea (Gastrointestinal disorders) | 3 (3) — One event in one affected subject was determined to be related to HepQuant SHUNT Liver Diagnostic Kit
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Related to HepQuant SHUNT Liver Diagnostic Kit
Flushing (Vascular disorders) | 1 (1) — Related to HepQuant SHUNT Liver Diagnostic Kit
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 3 (5)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Corona virus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Eye pain (Eye disorders) | 1 (1)
Food allergy (Immune system disorders) | 1 (1)
Coronavirus test positive (Investigations) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03583996/Prot_SAP_000.pdf